CLINICAL TRIAL: NCT03302767
Title: CAP'Onco : Psychological and Social Consultation of Professional Accompaniment in Oncology
Acronym: CAP'ONCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IB2017-03; 2017-A01251-52 (Other: ANSM)
Record Dates: First submitted 2017-05-12; First posted 2017-10-05 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Cancer
Keywords: Oncology; Work Keeping; Social difficulties; Cognitive Disorders
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological and Social Consultation (Experimental): Psychological and Social Consultation
  Interventions: Other: Psychological and Social Consultation

INTERVENTIONS:
Other: Psychological and Social Consultation — Psychological and Social Consultation at Baseline, during the study and at the end of follow-up

SUMMARY:
This patient support system is designed to help patients regain their professional activity after their treatment. It's a 3-Axis neuropsycho-social synergy on 3 axes:

* A weekly pluridisciplinary consultation in tandem (Social worker + Psychologist / Neuropsychologist)
* Monthly information meetings and workshops (TIC'Onco reunions: collective information times and Cogit'Onco workshops: cognitive workshops
* An information booklet "Prepare the work return" The aim of this research is to evaluate efficiency in term of quality of life improvement linked to work status, utility, feasibility and patients' satisfaction.

The aim of this research is to evaluate efficiency in term of quality of life improvement linked to work status, utility, feasibility and patients' satisfaction.

DETAILED DESCRIPTION:
Unmet need characterize in 4 points:

* Cancer and survival: challenges for cancer patients who want to work while being treated
* Cancer and career: Job instability for cancer patients
* Difficulties and isolation of patients due to a lack of coordination between healthcare professionals and colleagues/management
* Post-treatment cognitive troubles stress and hindered patient return to employment: chemo brain This research-action will propose and evaluate a concrete device: To maintain a professional activity with the support of CAP'Onco during treatment, to balance between quality of life, managing the "cancer event" and the psychosocial consequences for professional experience, to provide an early, durable and multimodal support to improve work keeping and anticipate return to employment

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Institut Bergonié
* Informed Consent signed.
* Patients affiliated to a French social
* living in Gironde
* Professional activity at the time of diagnosis
* Treated for - breast cancer, Hodgkin's or non-Hodgkin's lymphoma (non-cerebral), testicular cancer
* CURATIVE support
* At any time during treatment (chemotherapy or radiotherapy, or immunotherapy)

Exclusion Criteria:

* Patient deprived of liberty or subject to a legal protection measure
* History of cancers
* Cerebral pathology and / or brain metastasis

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique GERAT-MULLER, PhD, Principal Investigator — Institut Bergonié - Supportive Oncology Care
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychological and Social Consultation
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Psychological and Social Consultation
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 44.9 [31.2 to 55.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 29
Marital Status [Count of Participants; unit: Participants]
  Married | 11
  As a couple | 7
  Single | 10
  Widower | 1
SOCIO-PROFESSIONAL CATEGORY [Count of Participants; unit: Participants]
  craftsman, shopkeeper, business owner | 3
  executive, intellectual profession | 6
  intermediate profession | 5
  employee | 14
  person without professional activity | 1
PROFESSIONAL STATUS [Count of Participants; unit: Participants]
  Public Sector | 13
  Private Sector | 12
  Self-employed worker | 3
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life : EORTC QLQ-C30 Scores
Description: Standardised QLQ-C30 scoring according to EORTC scoring manual (Fayers et al. EORTC QLQ-C30 scoring manual. 2001).
  15 dimensions are presented below. Each dimension is a standardised score ranges from 0 to 100. A low score corresponds to a low functional level, an absence of symptoms or a low level of QoL/ overall health and, conversely, so that a high score corresponds to a high functional level, a high presence of symptoms or a high level of QoL/overall health.
Time Frame: At baseline and 5 months
Population: * At baseline, 1 patient did not complete the QLQ-C30 questionnaire. And of the remaining 28 patients, 1 patient has missing data for the score 'Dyspnoea'.
  * At 5 months, 1 patient did not complete the QLQ-C30 questionnaire. And of the remaining 28 patients :
    * 1 patient has missing data for the scores 'Constipation' and 'Diarrhoea'
    * 1 another patient has missing data for the score 'Fatigue'
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Psychological and Social Consultation
Number analyzed (Participants) | 29
scores on a scale
  Global health status/ quality of life - Baseline: number analyzed (Participants) | 28
  Global health status/ quality of life - Baseline | 61.0 [54.3 to 67.7]
  Global health status/ quality of life - 5 months | 70.8 [66.1 to 75.5]
  Physical functioning - Baseline: number analyzed (Participants) | 28
  Physical functioning - Baseline | 82.9 [78.8 to 86.9]
  Physical functioning - 5 months | 83.2 [78.7 to 87.6]
  Role functioning - Baseline: number analyzed (Participants) | 28
  Role functioning - Baseline | 72.6 [63.6 to 81.6]
  Role functioning - 5 months | 78.6 [70.2 to 87.0]
  Emotional functioning - Baseline: number analyzed (Participants) | 28
  Emotional functioning - Baseline | 61.0 [51.3 to 70.7]
  Emotional functioning - 5 months | 67.0 [57.9 to 76.0]
  Cognitive functioning - Baseline: number analyzed (Participants) | 28
  Cognitive functioning - Baseline | 61.3 [52.7 to 69.9]
  Cognitive functioning - 5 months | 73.2 [65.1 to 81.3]
  Social functioning - Baseline: number analyzed (Participants) | 28
  Social functioning - Baseline | 73.2 [62.9 to 83.5]
  Social functioning - 5 months | 82.1 [73.9 to 90.4]
  Fatigue - Baseline: number analyzed (Participants) | 28
  Fatigue - Baseline | 47.6 [40.0 to 55.2]
  Fatigue - 5 months | 43.6 [35.3 to 52.0]
  Nausea/ vomiting - Baseline: number analyzed (Participants) | 28
  Nausea/ vomiting - Baseline | 3.6 [0.3 to 6.8]
  Nausea/ vomiting - 5 months | 3.0 [-0.1 to 6.0]
  Pain - Baseline: number analyzed (Participants) | 28
  Pain - Baseline | 38.7 [29.5 to 47.8]
  Pain - 5 months | 33.3 [23.2 to 43.4]
  Dyspnoea - Baseline: number analyzed (Participants) | 27
  Dyspnoea - Baseline | 24.7 [14.0 to 35.4]
  Dyspnoea - 5 months | 16.7 [8.4 to 24.9]
  Insomnia - Baseline: number analyzed (Participants) | 28
  Insomnia - Baseline | 52.4 [38.1 to 66.6]
  Insomnia - 5 months | 41.7 [29.2 to 54.2]
  Appetite loss - Baseline: number analyzed (Participants) | 28
  Appetite loss - Baseline | 9.5 [3.6 to 15.5]
  Appetite loss - 5 months | 6.0 [0.9 to 11.0]
  Constipation - Baseline: number analyzed (Participants) | 28
  Constipation - Baseline | 21.4 [12.0 to 30.9]
  Constipation - 5 months | 16.0 [3.7 to 28.4]
  Diarrhoea - Baseline: number analyzed (Participants) | 28
  Diarrhoea - Baseline | 8.3 [1.6 to 15.0]
  Diarrhoea - 5 months | 3.7 [-1.9 to 9.3]
  Financial difficulties - Baseline: number analyzed (Participants) | 28
  Financial difficulties - Baseline | 21.4 [11.3 to 31.5]
  Financial difficulties - 5 months | 15.5 [6.5 to 24.4]

2. Primary Outcome: Cognitive Complaints : FACT Cog Scale Scores
Description: Cognitive complaints were evaluated by using the french Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) scale version 3
  Assessed using median total score (range 0-132) and median scores of these 4 dimensions :
  * Perceived Cognitive Impairment (range 0-72)
  * Impact on quality of life (range 0-16)
  * Comments from others (range 0-16)
  * Perceived Cognitive Skills (range 0-28) Higher scores indicate better cognitive functioning.
Time Frame: At baseline and 5 months
Population: * At baseline, 2 patients did not complete the Cognitive complaints questionnaire
  * At 5 months, 1 patient did not complete the Cognitive complaints questionnaire
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Psychological and Social Consultation
Number analyzed (Participants) | 29
scores on a scale
  Perceived Cognitive Impairment - Baseline: number analyzed (Participants) | 27
  Perceived Cognitive Impairment - Baseline | 39 [8 to 69]
  Perceived Cognitive Impairment - 5 months: number analyzed (Participants) | 28
  Perceived Cognitive Impairment - 5 months | 50.5 [7 to 72]
  Impact on quality of life - Baseline: number analyzed (Participants) | 27
  Impact on quality of life - Baseline | 8 [0 to 16]
  Impact on quality of life - 5 months: number analyzed (Participants) | 28
  Impact on quality of life - 5 months | 14.0 [0 to 16]
  Comments from others - Baseline: number analyzed (Participants) | 27
  Comments from others - Baseline | 15 [5 to 16]
  Comments from others - 5 months: number analyzed (Participants) | 28
  Comments from others - 5 months | 16 [3 to 16]
  Perceived Cognitive Skills - Baseline: number analyzed (Participants) | 27
  Perceived Cognitive Skills - Baseline | 13 [3 to 25]
  Perceived Cognitive Skills - 5 months: number analyzed (Participants) | 28
  Perceived Cognitive Skills - 5 months | 17.5 [0 to 27]
  Total score - Baseline: number analyzed (Participants) | 27
  Total score - Baseline | 75 [16 to 125]
  Total score - 5 months: number analyzed (Participants) | 28
  Total score - 5 months | 96 [33 to 127]

3. Primary Outcome: Professional Recovery Scale Scores
Description: Professional recovery was evaluated by using the Scale of motivation to Professional recovery.
  This scale was constructed for the needs of this exploratory research and has for vocation a later validation.
  It includes 62 questions and was assessed using median scores of these 7 dimensions :
  * Work and administrative process (0-100)
  * Positioning in relation to the job-post-mission (0-100)
  * Emotion and work (0-100)
  * Labour relations (0-100)
  * Work and physical/intellectual conditions (0-100)
  * Privacy and work (0-100)
  * Return to work (0-20) Higher scores represent better outcomes
Time Frame: At baseline and 5 months
Population: * At baseline, 1 patient did not complete the Professional recovery questionnaire
  * At 5 months :
    * 3 patients have missing data for the scores 'Work and administrative process', 'Work and physical/intellectual conditions' and 'Privacy and work'
    * 4 patients have missing data for the scores 'Positioning in relation to the job-post-mission', 'Emotion and work' and 'Labour relations'
    * 1 patient has missing data for the score 'Return to work'
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Psychological and Social Consultation
Number analyzed (Participants) | 29
scores on a scale
  Work and administrative process - Baseline: number analyzed (Participants) | 28
  Work and administrative process - Baseline | 58 [44 to 73]
  Work and administrative process - 5 months: number analyzed (Participants) | 26
  Work and administrative process - 5 months | 61 [34 to 80]
  Positioning in relation to the job-post-mission - Baseline: number analyzed (Participants) | 28
  Positioning in relation to the job-post-mission - Baseline | 40.5 [13 to 75]
  Positioning in relation to the job-post-mission - 5 months: number analyzed (Participants) | 25
  Positioning in relation to the job-post-mission - 5 months | 50 [10 to 73]
  Emotion and work - Baseline: number analyzed (Participants) | 28
  Emotion and work - Baseline | 58.5 [28 to 88]
  Emotion and work - 5 months: number analyzed (Participants) | 25
  Emotion and work - 5 months | 60 [33 to 91]
  Labour relations - Baseline: number analyzed (Participants) | 28
  Labour relations - Baseline | 55 [11 to 90]
  Labour relations - 5 months: number analyzed (Participants) | 25
  Labour relations - 5 months | 59 [28 to 90]
  Work and physical/intellectual conditions - Baseline: number analyzed (Participants) | 28
  Work and physical/intellectual conditions - Baseline | 42 [17 to 88]
  Work and physical/intellectual conditions - 5 months: number analyzed (Participants) | 26
  Work and physical/intellectual conditions - 5 months | 52.5 [28 to 84]
  Privacy and work - Baseline: number analyzed (Participants) | 28
  Privacy and work - Baseline | 50.5 [29 to 72]
  Privacy and work - 5 months: number analyzed (Participants) | 26
  Privacy and work - 5 months | 60.5 [25 to 77]
  Return to work - Baseline: number analyzed (Participants) | 28
  Return to work - Baseline | 10 [1 to 20]
  Return to work - 5 months: number analyzed (Participants) | 28
  Return to work - 5 months | 14 [2 to 20]

4. Secondary Outcome: Tiredness : Piper MFI-20 Scale Scores
Description: Tiredness was evaluated by using the Piper Multidimensional Fatigue Inventory (MFI-20) revised scale
  Assessed using median total score (range 0-10) and median scores of these 4 tiredness dimensions :
  * Behavioural
  * Emotional
  * Sensory
  * Cognitive-mood Each dimension has range 0-10 with following interpretation: higher scores indicate greater severity of fatigue
Time Frame: At baseline and 5 months
Population: * At baseline:
    * 2 patients have missing data for the scores 'Emotional dimension', Behavioural dimension' and 'Sensory dimension'
    * 3 patients have missing data for the score 'Cognitive-mood dimension'
    * 3 patients finally have missing data for 'Total Score Fatigue Scale'
  * At 5 months, 1 patient did not complete the Tiredness questionnaire
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Psychological and Social Consultation
Number analyzed (Participants) | 29
scores on a scale
  Emotional dimension - Baseline: number analyzed (Participants) | 27
  Emotional dimension - Baseline | 5.4 [1.6 to 9.8]
  Behavioural dimension - 5 months: number analyzed (Participants) | 28
  Behavioural dimension - 5 months | 4.7 [0.5 to 9.2]
  Behavioural dimension - Baseline: number analyzed (Participants) | 27
  Behavioural dimension - Baseline | 5.3 [0.0 to 9.7]
  Emotional dimension - 5 months: number analyzed (Participants) | 28
  Emotional dimension - 5 months | 5.7 [2.0 to 9.8]
  Sensory dimension - Baseline: number analyzed (Participants) | 27
  Sensory dimension - Baseline | 4.2 [0.6 to 7.6]
  Sensory dimension - 5 months: number analyzed (Participants) | 28
  Sensory dimension - 5 months | 4.0 [0.8 to 7.2]
  Cognitive-mood dimension - Baseline: number analyzed (Participants) | 26
  Cognitive-mood dimension - Baseline | 4.8 [0.5 to 7.7]
  Cognitive-mood dimension - 5 months: number analyzed (Participants) | 28
  Cognitive-mood dimension - 5 months | 3.9 [0.3 to 6.3]
  Total Score Fatigue Scale - Baseline: number analyzed (Participants) | 26
  Total Score Fatigue Scale - Baseline | 5.2 [0.9 to 7.8]
  Total Score Fatigue Scale - 5 months: number analyzed (Participants) | 28
  Total Score Fatigue Scale - 5 months | 4.7 [1.5 to 6.5]

5. Secondary Outcome: Anxio-depressive Troubles : HAD Scale Scores
Description: Anxio-depressive troubles were evaluated by using the Hospital Anxiety and Depression (HAD) scale.
  Assessed using median scores of these 2 dimensions :
  * Anxiety
  * Depression Each dimension has range 0-21 with following interpretation: higher scores represent worse outcomes (0-7 normal; 8-10 mild; 11-14 moderate; 15-21 severe)
Time Frame: At baseline and 5 months
Population: * At baseline, 2 patients did not complete the Anxio-depressive troubles questionnaire
  * At 5 months ,1 patient did not complete the Anxio-depressive troubles questionnaire
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Psychological and Social Consultation
Number analyzed (Participants) | 29
scores on a scale
  Anxiety score - Baseline: number analyzed (Participants) | 27
  Anxiety score - Baseline | 10.0 [1 to 19]
  Anxiety score - 5 months: number analyzed (Participants) | 28
  Anxiety score - 5 months | 8 [2 to 18]
  Depression score - Baseline: number analyzed (Participants) | 27
  Depression score - Baseline | 7.0 [4 to 18]
  Depression score - 5 months: number analyzed (Participants) | 28
  Depression score - 5 months | 6.5 [3 to 12]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed (so Total Number At Risk = 0).
Arm/Group | Psychological and Social Consultation
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT03302767/Prot_SAP_000.pdf